CLINICAL TRIAL: NCT06977789
Title: Comparison of Holter vs S-Patch for Arrhythmia Detection in Older Falls Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Changi General Hospital (Other)
Collaborators: Samsung SDS Asia Pacific Pte Ltd (Unknown)
Responsible Party: Principal Investigator, Colin Yeo, Senior Consultant, Changi General Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 2019/2960
Record Dates: First submitted 2025-04-29; First posted 2025-05-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Bradyarrhythmia; Arrythmia
MeSH Terms: conditions — Bradycardia; Arrhythmias, Cardiac | interventions — Electrocardiography, Ambulatory

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Holter for 24 hour follow by S Patch3-Cardio/S-Patch Ex for 72 hours) (Active Comparator): Holter for 24 hour follow by S Patch3-Cardio/S-Patch Ex for 72 hours
  Interventions: Device: S Patch3-Cardio/S-Patch Ex; Device: Holter
- Group B (S Patch3-Cardio/S-Patch Ex for 72 hours follow by Holter for 24hour). (Active Comparator): S Patch3-Cardio/S-Patch Ex for 72 hours follow by Holter for 24hour
  Interventions: Device: S Patch3-Cardio/S-Patch Ex; Device: Holter

INTERVENTIONS:
Device: S Patch3-Cardio/S-Patch Ex — S Patch3-Cardio/S-Patch Ex for 72 hours
Device: Holter — Holter for 24 hours

SUMMARY:
The aim of this study is to compare Holter versus S patch in a group of elderly patients who are referred to the Geriatrics service in Changi General Hospital for falls from Accident and Emergency department, clinic and wards.

The investigator hope to assess the feasibility, adherence and patient acceptability as an alternative to Holter monitoring. The investigator also hope to learn if S-Patch EX monitoring system can be as effective or equivalent to Holter in the monitoring of arrhythmias and the possibility of deploying it for longer term monitoring of arrhythmias.

Participants who consented to be in this study will be offered S patch and Holter consecutively. Holter will be worn for 24 hours and S patch will be worn for 72 hours. The order which Holter or S patch will be worn first will be determined via randomisation.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 60 to 120 year old inclusive
2. Refer for Holter testing as part of clinical care
3. Participants with symptoms suspected to be due to bradyarrhythmia. This could include, but not limited to unwitnessed fall, syncope, near syncope.

Exclusion Criteria:

1. Participants who are already known to have significant bradyarrhythmia who would benefit from a permanent pacemaker.
2. Patients unable to tolerate Holter monitoring.

Ages: 60 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2020-07-03 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-12-25 (Actual)

PRIMARY OUTCOMES:
Participant's Compliance | From date of randomization until the day participant completed both device monitoring, assessed up to 4 days.
  An events diary and questionnaire to evaluate their preference between Holter and the S-Patch recorder. The hours of recording from both devices will also be captured in both devices report.

SECONDARY OUTCOMES:
Device sensitivity and specificity | 72 hours for S Patch3-Cardio/S-Patch Ex and 24hours for Holter
  Assess sensitivity and specificity of S Patch3-Cardio/S-Patch Ex compared to Holter to diagnose the bradyarrhythmia/arrhythmia. The sensitivity and specificity will be analyzed from the device report. Outcome comparison between the two treatment arms using McNemars test.
Durability of the device | 72 hours for S Patch3-Cardio/S-Patch Ex and 24hours for Holter
  Durability of the device in longer term monitoring and in real world situation. The hours of monitoring from S Patch3-Cardio/S-Patch Ex is compare with hours of monitoring from Holter to see if 72 hours of monitoring will have a better outcome compare to only 24hrs of recording. The duration of recording are taken from the device monitoring reports.

CONTACTS AND LOCATIONS:
Overall Officials: Yeo Colin, Principal Investigator — Changi General Hospital
Locations (1):
- Changi General Hospital, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No